CLINICAL TRIAL: NCT03539224
Title: Antiretroviral Treatment Guided by Proviral Genotype: Pilot Trial of Proof of Concept.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto de Investigación Hospital Universitario La Paz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ART-PRO; 2017-000151-10 (EudraCT Number)
Record Dates: First submitted 2018-04-02; First posted 2018-05-29 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Intervention Model Description: Single arm opened with Intervention Type of Drug: Dolutegravir (DTG) and Lamivudina (3TC)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dolutegravir (DTG) + Lamivudine (3TC) (Experimental): Eligible subjects will receive one 50 mg tablet of DTG plus 300 mg 3TC tablet orally once daily upto 48 weeks
  Interventions: Drug: Dolutegravir (DTG); Drug: Lamivudine (3TC)

INTERVENTIONS:
Drug: Dolutegravir (DTG) — DTG 50 mg tablet will be orally administered once daily with or without food upto 48 weeks
  Other Names: Tivicay
Drug: Lamivudine (3TC) — Lamivudine will be dispensed as 300 mg white, diamond shaped, scored, film coated tablets. It will be orally administered once daily with or without food upto 48 weeks.
  Other Names: Epivir

SUMMARY:
Phase IIa, open clinical trial, pilot, single arm and proof of concept.

DETAILED DESCRIPTION:
Proof of concept trial evaluating safety and efficacy of treatment with Dolutegravir (DTG) + lamivudine (3TC) once daily in suppressed participants with history of previous treatment with 3TC or emtricitabine (FTC). Half of the participants will have history of failure with 3TC or FTC and M184V/I or K65R/E/N mutations in previous plasma genotypes, although to be eligible these mutations cannot be detectable at study entry in proviral DNA.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 infected patients.
2. Age> 18 years.
3. Receiving stable antiretroviral treatment for at least 3 months.
4. Current or historical treatment with 3TC or FTC.
5. Willing to change antiretroviral treatment due to intolerance or interest in simplification.
6. Undetectable viral load (<50 cop/mL) for at least 1 year prior to the inclusion. A single viral load >50cop/ml (≤500 copies/ml) is allowed before the three months prior to inclusion in the study, preceded and followed by an undetectable determination.
7. Current level of CD4> 350 cells/μL.
8. Naïve to integrase inhibitors.
9. Patient able to understand and give written informed consent.
10. For those included in group 1 (20 patients): No previous history of virological failure with ART regimen that included 3TC or FTC or previous virological failure had a population genotype without M184V/I or K65R/E/N mutations.
11. For those included in group 2 (20 patients): previous history of virological failure with ART regimen that included 3TC or FTC and historical genotype with M184V/I or K65R/E/N mutations.

Exclusion Criteria:

1. Detection of any of the following mutations in proviral DNA in peripheral blood by conventional sequencing: M184V/I or K65R/E/N.
2. Pregnant, lactating or child-bearing women who do not commit to using an adequate contraceptive method.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with undetectable viral load (<50 copies / mL) at 48 weeks | Week 48
  - Efficacy: Proportion of patients with undetectable viral load (<50 copies / mL) at 48 weeks of follow-up, according to the FDA snapshot algorithm in the population "by intention to treat-exposed". The intention-to-treat population includes all patients who have received at least one dose of DTG and 3TC.

SECONDARY OUTCOMES:
Proportion of patients with virological failure at 24 weeks | Week 24
  Proportion of patients with viral load <50 copies/ml at week 24, according to the FDA snapshot algorithm in the population "by intention to treat-exposed".
Proportion of patients with virological failure at 48 weeks | Week 48
  Proportion of patients with virological failure at week 48 according to the FDA snapshot algorithm.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Since baseline visits to week 48
  Incidence of adverse events and discontinuation of treatment due to toxicity or intolerance.
Evaluation of the appearance of genotypic resistance mutations (1) | Week 48
  Incidence of genotypic resistance mutations in patients with virological failure at week 48. Description and frequency of genotypic resistance mutations.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

REFERENCES:
- [Derived] De Miguel Buckley R, Rial-Crestelo D, Montejano R, Pinto A, Jimenez-Gonzalez M, Lagarde M, Esteban-Cantos A, Aranguren-Rivas P, Cadinanos J, Bisbal O, Castro JM, Santacreu-Guerrero M, Bermejo-Plaza L, Moreno V, Hernando A, Martin-Carbonero L, Rubio R, Delgado R, Arribas JR, Pulido F; Antiretroviral Treatment Guided by Proviral Genotype (ART-PRO) Study Group. Long-term Evaluation of Residual Viremia in a Clinical Trial of Dolutegravir Plus Lamivudine as Maintenance Treatment for Participants With and Without Prior Lamivudine Resistance. Open Forum Infect Dis. 2022 Nov 8;9(11):ofac610. doi: 10.1093/ofid/ofac610. eCollection 2022 Nov. PMID 36447613
- [Derived] De Miguel R, Rial-Crestelo D, Dominguez-Dominguez L, Montejano R, Esteban-Cantos A, Aranguren-Rivas P, Stella-Ascariz N, Bisbal O, Bermejo-Plaza L, Garcia-Alvarez M, Alejos B, Hernando A, Santacreu-Guerrero M, Cadinanos J, Mayoral M, Castro JM, Moreno V, Martin-Carbonero L, Delgado R, Rubio R, Pulido F, Arribas JR; ART-PRO, PI16/00837-PI16/00678 study group. Dolutegravir plus lamivudine for maintenance of HIV viral suppression in adults with and without historical resistance to lamivudine: 48-week results of a non-randomized, pilot clinical trial (ART-PRO). EBioMedicine. 2020 May;55:102779. doi: 10.1016/j.ebiom.2020.102779. Epub 2020 May 11. PMID 32408111